CLINICAL TRIAL: NCT01274572
Title: Blood Samples to Evaluate Immune Response to Provenge® (Sipuleucel-T) inHormone Refractory Metastatic Prostate Cancer Patients
Brief Title: Blood for Immune Response to Provenge® in HRPC
Status: Withdrawn | Type: Observational
Why Stopped: Drug became available with insurance reimbursement
Sponsor: Mary Crowley Medical Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: MC 10-11
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is being conducted to assess and monitor immune response in patients with minimally symptomatic or asymptomatic hormone refractory prostate cancer who will be receiving Provenge® (Sipuleucel-T) therapy as part of their standard of care treatment regimen.

DETAILED DESCRIPTION:
This study is being conducted to assess and monitor immune response in patients with minimally symptomatic or asymptomatic hormone refractory prostate cancer who will be receiving Provenge® (Sipuleucel-T) therapy as part of their standard of care treatment regimen. The trial only involves the collection of additional blood samples for the purposes of monitoring immune response. These samples will be taken at 7 time points before, during and after patients receive Provenge® (Sipuleucel-T). There will be no other study-specific procedures performed (other than the blood draws) nor any use of investigational agents in this study.

ELIGIBILITY:
Inclusion Criteria:

Patients who plan to receive standard of care Provenge® (Sipuleucel-T) at their primary physican's office.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects that will be included in this study will be receiving Provenge as standard of care treatment for their prostate cancer and will be willing to consent to the additional blood draws.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Immune Response | Additional Blood Sample
  Standard of Care Drug Immune Response

CONTACTS AND LOCATIONS:
Overall Officials: John Nemunaitis, MD, Principal Investigator — Mary Crowley Cancer Research Centers